CLINICAL TRIAL: NCT07134075
Title: Safety and Efficacy of Intracochlear Injection of Glucocorticoid Through the Round Window Membrane in Patients With Total Sudden Sensorineural Hearing Loss
Brief Title: Intracochlear Injection of Glucocorticoid
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: intracochlear glucocorticoid; 82225014 (Other Grant/Funding Number: National Science Foundation of China)
Record Dates: First submitted 2025-07-30; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sudden Sensorineural Hearing Loss (SSNHL)
Keywords: intracochlear injection; glucocorticoid
MeSH Terms: conditions — Hearing Loss, Sudden

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: single blinded (participant and outcomes assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: intracochlear triamcinolone acetonide injection (Experimental): intracochlear injection of triamcinolone acetonide through the round window membrane
  Interventions: Drug: intracochlear triamcinolone acetonide injection
- Group B: intracochlear dexamethasone injection (Experimental): intracochlear injection of dexamethasone through the round window membrane
  Interventions: Drug: intracochlear injection of dexamethasone through the round window membrane
- Group C: intracochlear dexamethasone injection and intratympanic dexamethasone injection (Experimental): intracochlear injection of dexamethasone through the round window membrane and intratympanic dexamethasone injection through the tympanic membrane
  Interventions: Drug: intracochlear dexamethasone injection and intratympanic dexamethasone injection
- Group D: intratympanic dexamethasone injection (Active Comparator): intratympanic dexamethasone injection tympanic membrane，once every other day, for a total of 4 injections.
  Interventions: Drug: intratympanic dexamethasone injection

INTERVENTIONS:
Drug: intracochlear triamcinolone acetonide injection — intracochlear triamcinolone acetonide injection of through the round window membrane
  Other Names: intracochlear triamcinolone acetonide （40mg/ml, 30μl）injection
  Arms: Group A: intracochlear triamcinolone acetonide injection
Drug: intracochlear injection of dexamethasone through the round window membrane — intracochlear injection of dexamethasone sodium phosphate through the round window membrane
  Other Names: intracochlear injection of dexamethasone sodium phosphate（7.5mg/ml, 30μl）through the round window membrane
  Arms: Group B: intracochlear dexamethasone injection
Drug: intracochlear dexamethasone injection and intratympanic dexamethasone injection — intracochlear dexamethasone sodium phosphate injection of through the round window membrane, intratympanic dexamethasone sodium phosphate injection through the tympanic membrane
  Other Names: intracochlear injection of dexamethasone sodium phosphate through the round window membrane (7.5mg/ml, 30μl) and intratympanic dexamethasone sodium phosphate injection (10mg/ml)
  Arms: Group C: intracochlear dexamethasone injection and intratympanic dexamethasone injection
Drug: intratympanic dexamethasone injection — intratympanic dexamethasone sodium phosphate injection (10mg/ml) through tympanic membrane，once every other day, for a total of 4 injections.
  Other Names: intratympanic dexamethasone sodium phosphate injection (10mg/ml)
  Arms: Group D: intratympanic dexamethasone injection

SUMMARY:
This study is a prospective, randomized pilot study. To verify safety and efficacy of intracochlear injection of glucocorticoid through the round window membrane in patients with total sudden sensorineural hearing loss safety and efficacy in total sudden sensorineural hearing loss patients as an early salvage therapy.

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. Whether is it safe when total sudden sensorineural hearing loss patients receive intracochlear injection of glucocorticoid through the round window membrane.
2. Whether is it effective in reversing hearing capability when total sudden sensorineural hearing loss patients receive intracochlear injection of glucocorticoid through the round window membrane.
3. Whether is intracochlear glucocorticoid injection more effective than intratympanic glucocorticoid injection for treating total sudden sensorineural hearing loss.
4. Which glucocorticoid intracochlear injection is more effective in patients with total sudden sensorineural hearing loss.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years Unilateral idiopathic sudden sensorineural hearing loss greater than 95dB at the average of 4 frequencies (500 Hz, 1000 Hz, 2000 Hz and 4000 Hz) in PTA (contralateral hearing is less than 30dB) at the onset of sudden hearing loss Participant who were treated with standard treatment for 14 days, but no recovery was confirmed as type IV (final hearing level with hearing gain of ≤15 dB) at the end of the 14-day treatment

Exclusion Criteria:

Bilateral sudden sensorineural hearing loss Hearing loss with known causes (e.g., Meniere's disease, retrocochlear pathology, history of otologic surgery, perilymphatic fistula, barotrauma) History in the past 6 months of ototoxic treatment such as chemotherapy, use of loop diuretics, high dose aspirin, etc History of sudden sensorineural hearing loss within the past 2 years History of ischemic diseases (cerebral infarction, myocardial infarction, peripheral arterial obstructive disease) Neuropsychiatric disorders (epilepsy, Parkinson's disease, Alzheimer's disease, multiple sclerosis) Severe hepatic or renal insufficiency The CT diagnosis is "abnormality of the round window niche"

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in pure tone audiometry (PTA) | Baseline, Week 2, Week 4, Week12, Week24
  hearing capacity of thresholds (PTA)
Change from Baseline in auditory brainstem response (ABR) | Baseline, Week 2, Week 4, Week12, Week24
  hearing capacity of thresholds (ABR)
Change from Baseline in auditory steady state response (ASSR) | Baseline, Week 2, Week 4, Week12, Week24
  hearing capacity of thresholds (ASSR)
Change from Baseline in speech Discrimination Scores | Baseline, Week 2, Week 4, Week12, Week24
  hearing capacity of thresholds (speech Discrimination Scores)

SECONDARY OUTCOMES:
change from baseline in tinnitus handicap inventory | Baseline, Week2, Week4, Week12, Week24
  The THI questionnaire includes functional, emotional, and catastrophic subscales. It consists of 25 questions. The total score is calculated by adding up the scores for all questions and classifying the severity of tinnitus as no handicap (0-16), mild handicap (18-36), moderate handicap (38-56), and severe handicap (58-100).
change from baseline in dizziness handicap inventory | Baseline, Week2, Week4, Week12, Week24
  The 25-item self-report Dizziness Handicap inventory (DHI) validated questionnaire that assesses functional, emotional and physical domains. Responses are graded 0 (no), 2 (sometimes) or 4 (yes) with higher scores indicating greater impact of dizziness maximum and maximum score of 100 points (15 minutes).
change from baseline in quality of life score | Baseline, Week2, Week4, Week12, Week24
  Quality of life questionnaire will be measured to compare the change in individual's health-related quality of life using face to face Interview for the scores. Higher scores mean better functioning or fewer symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Yilai Shu, MD, Ph.D, Principal Investigator — Eye & ENT Hospital, Fudan University, Shanghai, China
Locations (1):
- Fenyang Road 83, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The ethics committee may require approval for data sharing to ensure alignment with principles like beneficence and justice.

REFERENCES:
- [Background] Lv J, Wang H, Cheng X, Chen Y, Wang D, Zhang L, Cao Q, Tang H, Hu S, Gao K, Xun M, Wang J, Wang Z, Zhu B, Cui C, Gao Z, Guo L, Yu S, Jiang L, Yin Y, Zhang J, Chen B, Wang W, Chai R, Chen ZY, Li H, Shu Y. AAV1-hOTOF gene therapy for autosomal recessive deafness 9: a single-arm trial. Lancet. 2024 May 25;403(10441):2317-2325. doi: 10.1016/S0140-6736(23)02874-X. Epub 2024 Jan 24. PMID 38280389
- [Background] Choi JW, Lee CK, Kim SB, Lee DY, Ko SC, Park KH, Choi SJ. Potential benefits of salvage intratympanic dexamethasone injection in profound idiopathic sudden sensorineural hearing loss. Eur Arch Otorhinolaryngol. 2020 Aug;277(8):2219-2227. doi: 10.1007/s00405-020-05967-z. Epub 2020 Apr 15. PMID 32296977
- [Background] Plontke SK, Biegner T, Kammerer B, Delabar U, Salt AN. Dexamethasone concentration gradients along scala tympani after application to the round window membrane. Otol Neurotol. 2008 Apr;29(3):401-6. doi: 10.1097/MAO.0b013e318161aaae. PMID 18277312
- [Background] Matsui H, Lopez IA, Ishiyama G, Ishiyama A. Immunohistochemical localization of glucocorticoid receptors in the human cochlea. Brain Res. 2023 May 1;1806:148301. doi: 10.1016/j.brainres.2023.148301. Epub 2023 Mar 1. PMID 36868509
- [Background] Bird PA, Begg EJ, Zhang M, Keast AT, Murray DP, Balkany TJ. Intratympanic versus intravenous delivery of methylprednisolone to cochlear perilymph. Otol Neurotol. 2007 Dec;28(8):1124-30. doi: 10.1097/MAO.0b013e31815aee21. PMID 18043438
- [Background] Rauch SD, Halpin CF, Antonelli PJ, Babu S, Carey JP, Gantz BJ, Goebel JA, Hammerschlag PE, Harris JP, Isaacson B, Lee D, Linstrom CJ, Parnes LS, Shi H, Slattery WH, Telian SA, Vrabec JT, Reda DJ. Oral vs intratympanic corticosteroid therapy for idiopathic sudden sensorineural hearing loss: a randomized trial. JAMA. 2011 May 25;305(20):2071-9. doi: 10.1001/jama.2011.679. PMID 21610239
- [Background] Li W, Hartsock JJ, Dai C, Salt AN. Permeation Enhancers for Intratympanically-applied Drugs Studied Using Fluorescent Dexamethasone as a Marker. Otol Neurotol. 2018 Jun;39(5):639-647. doi: 10.1097/MAO.0000000000001786. PMID 29649043
- [Background] Silverstein H, Choo D, Rosenberg SI, Kuhn J, Seidman M, Stein I. Intratympanic steroid treatment of inner ear disease and tinnitus (preliminary report). Ear Nose Throat J. 1996 Aug;75(8):468-71, 474, 476 passim. PMID 8828271
- [Background] Wilson WR, Byl FM, Laird N. The efficacy of steroids in the treatment of idiopathic sudden hearing loss. A double-blind clinical study. Arch Otolaryngol. 1980 Dec;106(12):772-6. doi: 10.1001/archotol.1980.00790360050013. PMID 7002129
- [Background] McCabe BF. Autoimmune sensorineural hearing loss. Ann Otol Rhinol Laryngol. 1979 Sep-Oct;88(5 Pt 1):585-9. doi: 10.1177/000348947908800501. PMID 496191
- [Background] SCHUKNECHT HF. Ablation therapy in the management of Meniere's disease. Acta Otolaryngol Suppl. 1957;132:1-42. No abstract available. PMID 13457879
- [Background] Fishman JM, Cullen L. Investigating sudden hearing loss in adults. BMJ. 2018 Nov 12;363:k4347. doi: 10.1136/bmj.k4347. No abstract available. PMID 30420423
- [Background] Chandrasekhar SS, Tsai Do BS, Schwartz SR, Bontempo LJ, Faucett EA, Finestone SA, Hollingsworth DB, Kelley DM, Kmucha ST, Moonis G, Poling GL, Roberts JK, Stachler RJ, Zeitler DM, Corrigan MD, Nnacheta LC, Satterfield L, Monjur TM. Clinical Practice Guideline: Sudden Hearing Loss (Update) Executive Summary. Otolaryngol Head Neck Surg. 2019 Aug;161(2):195-210. doi: 10.1177/0194599819859883. PMID 31369349